CLINICAL TRIAL: NCT07009210
Title: Feasibility and Acceptability of AI Assisted Personalized Legacy Program (Reflections: My Story) for Patients With Serious Illness
Brief Title: AI Assisted Personalized Legacy Program (Reflections: My Story) for Patients With Serious Illness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Deirdre R. Pachman, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-008402
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Serious Illness; Existential Distress
Keywords: Legacy Work

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AI Assisted Personalized Legacy Program (Experimental)
  Interventions: Behavioral: AI Assisted Personalized Legacy Program

INTERVENTIONS:
Behavioral: AI Assisted Personalized Legacy Program — AI Assisted Personalized Legacy Program will be facilitated by a clinician trained in legacy work.

SUMMARY:
The purpose of this study is to determine if it is feasible and acceptable to recruit for and deliver the AI Assisted Personalized Legacy Program intervention to patients with serious illness.

DETAILED DESCRIPTION:
This study is an investigator-initiated, multi-site Mayo Clinic prospective minimal risk pilot study to determine feasibility and acceptability of an AI Assisted Personalized Legacy Program. The AI Assisted Personalized Legacy Program intervention is a brief, individualized psychotherapy that aims to relieve psycho-emotional and existential distress and improve the experiences of patients whose lives are impacted by serious illness. This therapy offers patients an opportunity to reflect on their life with a trained facilitator and share their thoughts and memories with family and other people in their life. The sessions are recorded and transcribed. The interventionist will work with patients to edit the document and provide a final legacy document for patient to keep and give to loved ones.

ELIGIBILITY:
Participant population: Adults with serious illness - defined as a health condition that carries a high risk of mortality

Inclusion Criteria for patients:

1. Age ≥18 years
2. English fluency
3. Provide informed consent
4. Ability to complete questionnaire(s) by themselves or with assistance

Exclusion Criteria:

1. Other psychological co-morbidities such as untreated schizophrenia, bipolar disease
2. Recent suicide attempt or psychiatric illness severe enough that hospitalization has been necessary in last 6 months
3. Active delirium
4. Advanced dementia
5. Participation in concurrent legacy offerings through the palliative care clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility Number | 2 years
  Study feasibility will be measured by the number of participants who enrolled and finished the study.
Acceptability | 5-10 days post-delivery of the final legacy document
  Acceptability, as measured by the 7-item Was it Worth It (WIWI Questionnaire).The questions are answered as either "yes, no, or uncertain," overall perception of quality of life change, overall perception of study experience, one open-ended feedback question, and an option to talk with someone about concerns. Positive responses indicate acceptability. Results are reported as individual items.

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Pachman, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials